Official Title: PET and MRI Brain Imaging of Bipolar Disorder

**NCT:** NCT01880957

**Document Date:** 11/14/2017

## Proposed Statistical Plan for [11C]-DASB (5-HTT) & [11C]-CUMI-101 (5-HT1A) from Parsey **Bipolar Study**

## **Outcomes**

**DASB:**  $V_T/f_p$  + bootstrap ROI error

**CUMI:** BP<sub>F</sub> + bootstrap ROI error (BP<sub>ND</sub>??)

#### A priori ROIs

DASB: acn, amy, midbrain, gcirc

CUMI: acn, amy, cin, dlPFC, parahippocampal gyrus, hippocampus, raphe

### **Statistical methods:**

Linear mixed models with subject fit as random variable LMM also with DASB & CUMI reference regions and fp

Key outcomes: p-values for main effects/interactions; overall model R<sup>2</sup> & p-value; standardized & unstandardized β's, 95% CIs, p-values for post-hocs

## **Covariates**

DASB: age

**CUMI**: age, sex, previous med status (dichotomous – w/n 4 years)

# Post-Treatment

Sample: HC, pre BPD, post BPD

**Question 1:** Do post-treatment BPD levels of DASB or CUMI differ from pre-treatment levels and HCs?

### Interactions of interest:

**Group** (relationship btw brain & Group across all regions) **Group\*ROI** (ROI-specific relationship btw brain & Group)

# Treatment Effects

Sample: pre/post BPD pairs

Tx response: % change in HDRS-24 (continuous) and remitter/non-remitter (dichotomous)

**Question 2:** Is the % change in DASB or CUMI associated with the treatment outcome?

## <u>Interactions of interest:</u>

**AHDRS** (relationship btw brain & Tx outcome across all regions) **ΔHDRS\*ROI** (ROI-specific relationship btw brain & Tx outcome)

#### **Dichotomous**

### Interactions of interest:

**Remission** (relationship btw brain & Tx outcome across all regions)

\_\_\_\_\_

# **Predicting Treatment Outcome**

Sample: pre BPD with pre HDRS-24 + >7-week HDRS-24

<u>Tx response:</u> % change in HDRS-24 (continuous) and remitter/non-remitter (dichotomous) (responder ??)

**Question 3:** Do pre DASB or CUMI in any of the *a prioris* predict treatment response? Are the *a prioris* independent predictors of treatment response?

#### Interactions of interest:

**PET roi** (pre-treatment PET in ROI predicts treatment response)

## <u>Interactions of interest:</u>

**PET\_roi** (any significant ROIs are independent predictors of Tx response (over and above the other ROIs))

Same models fit with dichotomous remission status

**Additional question:** Do pre DASB & CUMI together predict more of the variance in treatment response than either method alone?

Change in overall model R<sup>2</sup> from models with pre DASB & CUMI alone to combined model (If R<sup>2</sup> increases with both methods, tracers are predicting unique properties of Tx response)

**Question 4:** With what accuracy does pre DASB or CUMI predict treatment response?

Penalized logistic regression models

**Additional question:** With what accuracy do pre DASB & CUMI together predict treatment response Metrics of interest:

Accuracy, AUC, sensitivity, specificity, NPV, PPV, model factor importance ranking or % of variance explained with each factor